CLINICAL TRIAL: NCT06707714
Title: A Metabolomics-based Study to Explore the Mechanism of Remission of Metabolic Syndrome After Radical Gastrectomy
Acronym: Metabolomics
Status: Enrolling by invitation | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2511756041
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Syndrome; Gastric Cancer
Keywords: Gastric cancer; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Stomach Neoplasms | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Gastric cancer patients combine with hypertension: Gastric cancer patients diagnosed with hypertension
  Interventions: Diagnostic Test: hypertension
- Gastric cancer patients combine with diabetes: Gastric cancer patients diagnosed with diabetes
  Interventions: Diagnostic Test: diabetes
- Gastric cancer patients combine with fatty liver: Gastric cancer patients diagnosed with fatty liver
  Interventions: Diagnostic Test: fatty liver

INTERVENTIONS:
Diagnostic Test: hypertension — Gastric cancer patients with hypertension
  Groups: Gastric cancer patients combine with hypertension
Diagnostic Test: diabetes — diagnosed with diabetes
  Groups: Gastric cancer patients combine with diabetes
Diagnostic Test: fatty liver — diagnosed with fatty liver
  Groups: Gastric cancer patients combine with fatty liver

SUMMARY:
1. Analysis of preoperative and postoperative metabolite changes: Through metabolomics technology, the changes of preoperative and postoperative metabolites in patients with gastric cancer complicated with metabolic syndrome were systematically analyzed, and the key metabolites related to the remission of hypertension, hyperlipidemia, and diabetes after surgery were found.
2. Explore the influencing factors of postoperative remission of metabolic syndrome: Combined with clinical data, the association between various metabolites and the degree of postoperative remission was evaluated, and the main factors affecting postoperative remission were determined.
3. Reveal the mechanism of postoperative remission of metabolic syndrome: through multi-level metabolomics analysis, to clarify the metabolic pathways and mechanisms involved in the process of postoperative remission, and provide a new theoretical basis for the development of tumor metabolic surgery.

DETAILED DESCRIPTION:
This project will last 2-3 years. All patients who meet the inclusion and exclusion criteria will be divided into three groups according to the type of metabolic syndrome, including hypertension, diabetes and hyperlipidemia, with 50 cases in each group. Blood and feces of all patients were collected before surgery, 3 days after surgery, 6 months after surgery, and 1 year after surgery. The collected samples will be subjected to untargeted metabolomics analysis, using NMR-IVDr technology to detect the dynamic changes of all small molecular metabolites (mainly endogenous small molecular compounds with relative molecular weight within 1000 Da) in blood and feces before and after stimulation or disturbance without bias. The differential metabolites of blood glucose, blood lipid, cholesterol, insulin, renin, aldosterone, and angiotensin were screened by bioinformatics analysis, and the pathway analysis of differential metabolites was performed to reveal the potential physiological mechanism of postoperative hypertension, diabetes, and hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >18 years old. 2. Patients with hypertension or diabetes for more than 1 year before surgery. 3. Patients undergoing radical gastrectomy for gastric cancer.

Exclusion Criteria:

* 1. Gastric stump cancer. 2. Patients with distant metastasis. 3. Patients who underwent combined resection of other important organs. 4. Severe postoperative complications. 5. Patients who are using drugs that may significantly affect metabolic status (such as hormonal drugs, potent immunosuppressants, etc.). 6. Incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic disease remission | From date of surgery until the date of first documented postoperative complication, assessed up to 2 months after surgery.
  Metabolic disease remission was defined as any remission of hypertention, diabetes, or fatty liver measured 2 months after surgery. Hypertension remission was defined as arterial blood pressure less than 140/90 mmHg measured postoperatively in patients with preoperative comorbid hypertension. Diabetes remission was defined as fasting blood glucose less than 6 mmol/L measured postoperatively in patients with preoperative comorbid diabetes. Fatty liver remission was defined as liver function in the normal range measured by postoperative blood tests in patients with preoperative comorbid fatty liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The clinical sites of the experimental studies did not allow data sharing

REFERENCES:
- [Background] Cheng YX, Peng D, Tao W, Zhang W. Effect of oncometabolic surgery on gastric cancer: The remission of hypertension, type 2 diabetes mellitus, and beyond. World J Gastrointest Oncol. 2021 Sep 15;13(9):1157-1163. doi: 10.4251/wjgo.v13.i9.1157. PMID 34616520
- [Background] Nudotor RD, Prokopowicz G, Abbey EJ, Gonzalez A, Canner JK, Steele KE. Comparative Effectiveness of Roux-en Y Gastric Bypass Versus Vertical Sleeve Gastrectomy for Sustained Remission of Type 2 Diabetes Mellitus. J Surg Res. 2021 May;261:407-416. doi: 10.1016/j.jss.2020.12.024. Epub 2021 Jan 27. PMID 33515868
- [Background] Wang L, Hu D, Fan Z, Yu J, Zhang S, Lin Y, Chen X, Lin X, Yan X, Lin J, Peng F. Prognostic value of long-term antidiabetic and antihypertensive therapy in postoperative gastric cancer patients: the FIESTA study. BMC Gastroenterol. 2022 Oct 9;22(1):429. doi: 10.1186/s12876-022-02514-4. PMID 36210441
- [Background] Karimi P, Islami F, Anandasabapathy S, Freedman ND, Kamangar F. Gastric cancer: descriptive epidemiology, risk factors, screening, and prevention. Cancer Epidemiol Biomarkers Prev. 2014 May;23(5):700-13. doi: 10.1158/1055-9965.EPI-13-1057. Epub 2014 Mar 11. PMID 24618998